CLINICAL TRIAL: NCT01243333
Title: Multi-tracer PET Assessment of Response in Various Malignancies in Investigational and Recently Approved Therapeutic Agents
Brief Title: Multi-Tracer Positron Emission Tomography in Patients With Solid Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI43948; NCI-2011-03665 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-11-01; First posted 2010-11-18 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Fluorodeoxyglucose F18; alovudine; Magnetic Resonance Spectroscopy; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (multi-tracer PET scans) (Experimental): Patients undergo Positron Emission Tomography (PET) scans with [F-18]fluorodeoxyglucose and [F-18]fluorothymidine at baseline and within 7 days of completion of 1 or 2 (if the course is less than 3 weeks) therapeutic agent courses.
  Interventions: Radiation: [F-18]fluorodeoxyglucose; Radiation: [F-18]fluorothymidine; Procedure: Positron Emission Tomography; Radiation: Water O-15

INTERVENTIONS:
Radiation: [F-18]fluorodeoxyglucose — Undergo PET scans with [F-18]fluorodeoxyglucose
  Other Names: 18FDG; FDG; fludeoxyglucose F 18; Fludeoxyglucose F-18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Radiation: [F-18]fluorothymidine — Undergo PET scans with fluorine [F-18]fluorothymidine
  Other Names: 18F-FLT; 3'-Deoxy-3'-(18F) Fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; ALOVUDINE F-18; fluorothymidine F 18; FLT; Fluorothymidine F-18
Procedure: Positron Emission Tomography — Undergo PET scans with 3 radiotracers (fludeoxyglucose F 18, fluorine F 18 fluorothymidine, and water O-15)
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
Radiation: Water O-15 — Undergo PET scans with water O-15 tracers
  Other Names: [15O] Water; [15O]-H2O

SUMMARY:
This clinical trial studies multi-tracer positron emission tomography in patients with solid tumors. Diagnostic procedures, such as multi-tracer positron emission tomography, may help measure a patient's response to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Provide a reliable and validated cadre of positron emission tomography (PET) imaging derived biomarkers that yield a better understanding of: 1) early clinical benefit from various therapeutic agents in investigational and recently approved therapies; 2) efficacy during novel therapeutics in investigational therapeutics and recently approved therapeutics at Huntsman Cancer Institute (HCI); and 3) possible predict prognosis or other long-term outcomes.

II. Reveal a more detailed understanding of: (1) the in vivo biologic mechanisms of various therapeutic drugs in investigational therapies and recently approved therapies at HCI (2) information on why particular functional imaging profiles are seen in treated patients.

III. Reveal a more detailed understanding of how the combination of molecular imaging derived biomarkers will be potentially useful to physicians for decision making and for explanation of efficacy or outcomes for patients with cancer.

IV. Implement and evaluate a new imaging technology for multi-tracer PET imaging of these tracers.

OUTLINE:

Patients undergo PET scans with fludeoxyglucose (FDG) F 18 (18FDG), fluorine F 18 fluorothymidine (FLT), and water (H2O) O-15 (15O) tracers at baseline and within 7 days of completion of 1 or 2 (if the course is less than 3 weeks) therapeutic agent courses.

ELIGIBILITY:
Inclusion Criteria:

* Eligible adult patients currently meeting inclusion criteria and will be treated with an investigational or recently approved therapeutic agent at HCI; the patients must have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria; RECIST imaging must be current and have been obtained within 30 days prior to the baseline imaging session
* Patients must document their willingness to be followed for a period of time; for the purposes of imaging data analysis this will ideally be for at least 12 months after completing the investigational or recently approved therapy, however this may not always be possible; by signing informed consent, the patients are documenting their agreement to have clinical and radiographic endpoints and the results of histopathologic tissue analysis and other laboratory information entered into a research database
* All patients must sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines
* Female patients who are not postmenopausal or surgically sterile will undergo a serum pregnancy test prior to baseline and the subsequent set of multi-tracer PET scans; the serum pregnancy test must be performed within 48 hours prior to research PET imaging; a negative test will be necessary for such patients to undergo research PET imaging
* Serum glutamic oxaloacetic transaminase (SGOT) less than 4.0 times below or above the upper or lower limit range
* Serum glutamate pyruvate transaminase (SGPT) less than 4.0 times below or above the upper or lower limit range
* Alkaline phosphatase (ALK phos) less than 4.0 times below or above the upper or lower limit range
* Lactate dehydrogenase (LDH) less than 4.0 times below or above the upper or lower limit range
* Total bilirubin less than 4.0 times below or above the upper or lower limit range
* Serum electrolytes less than 4.0 times below or above the upper or lower limit range
* Complete blood count (CBC) with platelets less than 4.0 times below or above the upper or lower limit range
* Prothrombin time less than 2.5 times below or above the upper or lower limit range; for those patients receiving Coumadin or another anticoagulant the upper limit for prothrombin time must not exceed 6 times the upper limit of the normal range
* Partial thromboplastin time less than 2.5 times below or above the upper or lower limit range; for those patients receiving Coumadin or another anticoagulant the upper limit for partial thromboplastin time must not exceed 6 times the upper limit of the normal range
* Blood urea nitrogen (BUN) less than 4.0 times below or above the upper or lower limit range
* Creatinine less than 4.0 times below or above the upper or lower limit range
* Urinalysis less than 4.0 times below or above the upper or lower limit range; urinalysis abnormalities will not preclude the patient from being enrolled and studied

Exclusion Criteria:

* Patients with known allergic or hypersensitivity reactions to previously administered radiopharmaceuticals; patients with significant drug or other allergies or autoimmune diseases may be enrolled at the Investigator's discretion
* Patients who are pregnant or lactating or who suspect they might be pregnant; serum pregnancy tests will be obtained prior to the baseline and subsequent multi-tracer PET scans in female patients that are not postmenopausal or surgically sterile
* Adult patients who require monitored anesthesia for PET scanning
* Patients known to be human immunodeficiency virus (HIV) positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-02-02 (Actual); Primary Completion 2015-12-12 (Actual); Study Completion 2016-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Yap, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Multi-Tracer PET Scans: Patients undergo Positron Emission Tomography (PET) scans with [F-18]fluorodeoxyglucose and [F-18]fluorothymidine at baseline and within 7 days of completion of 1 or 2 (if the course is less than 3 weeks) therapeutic agent courses.
Period: Overall Study
Arm/Group | All Patients: Multi-Tracer PET Scans
Started | 26
Completed | 18
Not Completed | 8

BASELINE CHARACTERISTICS:
Groups:
- All Patients: Multi-Tracer PET Scans: Patients undergo PET scans with [F-18]fluorodeoxyglucose and [F-18]fluorothymidine at baseline and within 7 days of completion of 1 or 2 (if the course is less than 3 weeks) therapeutic agent courses.
Arm/Group | All Patients: Multi-Tracer PET Scans
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.08 (16.25)
Age, Continuous [Median (Full Range); unit: years] | 55 [25 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: FDG Therapeutic Response
Description: The patients underwent baseline and repeat PET/CT imaging (after one to two cycles of treatment) with [F-18]fluorodeoxyglucose (FDG) and [F-18]fluorothymidine (FLT). The percent change in the SUVmax for FDG was calculated and used to determine the response. Partial response (PR) was defined as 35% or greater reduction in SUVmax, Progressive Disease (PD) was defined as 35% or greater increase in SUVmax, and Stable Disease (SD) was defined as all other changes in SUVmax.
Time Frame: 1-2 cycles of treatment - approximately one month
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients: Multi-Tracer PET Scans
Number analyzed (Participants) | 18
Participants
  Partial Response (PR) | 10
  Stable Disease (SD) | 8
  Progressive Disease (PD) | 0

2. Primary Outcome: FLT Therapeutic Response
Description: The patients underwent baseline and repeat PET/CT imaging (after one to two cycles of treatment) with [F-18]fluorodeoxyglucose (FDG) and [F-18]fluorothymidine (FLT). The percent change in the SUVmax for FLT was calculated and used to determine the response. Partial response (PR) was defined as 35% or greater reduction in SUVmax, Progressive Disease (PD) was defined as 35% or greater increase in SUVmax, and Stable Disease (SD) was defined as all other changes in SUVmax.
Time Frame: 1-2 cycles of treatment - approximately one month
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients: Multi-Tracer PET Scans
Number analyzed (Participants) | 18
Participants
  Partial Response (PR) | 8
  Stable Disease (SD) | 8
  Progressive Disease (PD) | 2

3. Primary Outcome: Standard Therapeutic Response
Description: The patients underwent baseline and repeat PET/CT imaging (after one to two cycles of treatment) with [F-18]fluorodeoxyglucose (FDG) and [F-18]fluorothymidine (FLT). Percent change in lesion measurements according to standard response criteria for the patient's tumor type were obtained. For brain tumors, Response Assessment in Neuro-Oncology (RANO) criteria were used. Partial Response (PR) was defined as 50% or greater reduction in lesion measurements, Progressive Disease (PD) was 25% or greater increase in measurements, and Stable Disease (SD) was neither PD or PR. Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria were used for solid tumors, with PR defined as 30% or greater reduction in measurements, PD was 20% or greater increase in measurements, and SD was all other changes.
Time Frame: 1-2 cycles of treatment - approximately one month
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients: Multi-Tracer PET Scans
Number analyzed (Participants) | 18
Participants
  Partial Response (PR) | 4
  Stable Disease (SD) | 10
  Progressive Disease (PD) | 4

ADVERSE EVENTS:
Arm/Group | All Patients: Multi-Tracer PET Scans
All-Cause Mortality (participants affected / at risk) | 1/26
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients: Multi-Tracer PET Scans (N=26)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other: Death due to disease pr (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Death due to disease progression

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes